CLINICAL TRIAL: NCT03193710
Title: Comparison of the Effects of Total Intravenous Anesthesia and Inhalation Anesthesia on Lymphocytes in Patients Undergoing Colorectal Cancer Resection and the Mechanism Involved: a Single-center, Randomized, Prospective Study
Brief Title: The Effects of General Anesthetics on Lymphocytes in Patients Undergoing Colorectal Cancer Resection and Mechanism Involved
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guizhi Du (Other)
Responsible Party: Sponsor-Investigator, Guizhi Du, Associate Professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: WestChinaHospital
Record Dates: First submitted 2017-06-12; First posted 2017-06-21 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Cancer Metastatic; Survival Rate; General Anesthetics Toxicity; Lymphocyte Destruction; Molecular Mechanism of Pharmacological Action
Keywords: Intravenous anesthesia; Inhalational anesthesia; Colorectal cancer resection; Lymphocytes; Metastasis; Survival; Molecular mechanism
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Propofol; Sevoflurane; Remifentanil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood of the enrolled patients will be sampled at different time-points for examination of lymphocytes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Total intravenous anesthesia group: The anesthesia of patients in the total intravenous anesthesia group will be maintained with propofol and remifentanil.
  Interventions: Drug: Propofol; Drug: Remifentanil
- Inhalational anesthesia group: The anesthesia of patients in the inhalational anesthesia group will be maintained with sevoflurane and remifentanil.
  Interventions: Drug: Sevoflurane; Drug: Remifentanil

INTERVENTIONS:
Drug: Propofol — Propofol will be used for anesthesia maintenance in the total intravenous anesthesia group.
  Other Names: Diprivan
  Groups: Total intravenous anesthesia group
Drug: Sevoflurane — Sevoflurane will be used for anesthesia maintenance in the inhalation anesthesia group.
  Other Names: Abbvie
  Groups: Inhalational anesthesia group
Drug: Remifentanil — Remifentanil will be used for analgesia in both groups.
  Other Names: YiChang HumanWell Pharmaceutical Co.，LTD. China

SUMMARY:
The body immunity is important to the development of tumor. The immune system is in charge of monitoring and cleaning tumor cells in circulation. Anesthesia may alter the immune response and affect the elimination of tumor cells. The purpose of the trial is to test whether inhalational anesthetic is relevant to tumor metastasis and recurrence of patients undergoing colorectal cancer resection through depression of lymphocytes-mediated immunity.

DETAILED DESCRIPTION:
With the increasing number of patients diagnosed with colorectal cancer, the proportion of patients undergoing surgical resection with general anesthesia increased. However, the operation can lead tumor cells releasing into the blood or peritoneal implantation, and the impaired immune response can make patients susceptible to the development of tumor metastasis and recurrence which is the the main reason of death. It is well known that B lymphocytes and T lymphocytes are the main immune cells, and B lymphocytes by secreting antibodies are related to humoral immunity and T lymphocytes which play the most important role in antitumor are related to cell-mediated immunity. Surgery stress leads to metabolic and neuroendocrine changes causing significant depression of immunity. Although general anesthesia could reduce surgical stress, studies indicated general anesthetics including intravenous and inhalational agents both have variable effects on tumor cells growth by immuno-modulation and some cytokines. A number of studies have demonstrated deleterious effects on the function of lymphocytes associated with the administration of volatile inhalational anesthetic agents. It was suggested that the use of volatile inhalational agent may augment tumor cells growth by inhibiting the activity of lymphocytes, NK cells and dendritic cells which are important for recognizing, capturing and killing tumor cells, however, the alternative propofol has a converse (beneficial) effect by decreasing the plasma level of cytokines secreted by activated lymphocytes, macrophages and NK cells. The detailed mechanism of how volatile anesthetics affect the activity of antitumor cells remains unknown. Thus the investigators will conduct the clinical investigation to study the effect of volatile anesthetics on the immune response and metastasis in patients undergoing colorectal cancer resection, exploring molecular mechanism involved if inhalational anesthetics show an effect. The findings of this study would be valuable for anesthetic regimen guidance of colorectal cancer patients undergoing surgical resection in terms of long-term survival.

ELIGIBILITY:
Inclusion Criteria:

* All the patients diagnosed with colonal or rectal cancer
* Aged 18-65
* ASA I-III
* Assigned to receive resection surgery under general anesthesia, with an expected duration of 2 hours or more
* Agree to participate and give signed written informed consent.

Exclusion Criteria:

* Severe organic heart, liver and kidney diseases
* Diabetes or hemopoietic disorders
* Allergy to general anesthetics
* Family historical malignant hyperthermia
* Cognition dysfunction
* End-stage cancer or with over 2 cancer metastasis, pathological results were benign tumor or TNM stage was over T1- 3N0 - 2M0
* Other primary malignant tumor
* Immune deficiency or dysfunction or autoimmune disease or long-term usage of corticoids or immunosuppressants
* Receiving general anesthesia within the last 3 months before the resection surgery
* Perioperative transfusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colonal or rectal cancer undergoing cancer resection with general anesthesia
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline lymphocytes within postoperative 5 years | up to 5 years
  Blood will be drawn preoperatively ( at least 24 hours before surgery), prior to anesthesia induction, immediately postoperatively, 24 hours postoperatively, and at postoperative appointments for testing CD4+/CD8+, B lymphocytes, dendritic cells, natural killer cells
Cancer free survival | 5 years or as available
  Patients who remain alive without known colonal or rectal tumor recurrence

SECONDARY OUTCOMES:
Cancer recurrence rate | up to 5 years
  Patients who remain alive with known colonal or rectal tumor recurrence
Cancer metastasis rate | up to 5 years
  Patients who remain alive with known colonal or rectal tumor metastasis
Re-operation | up to 5 years
  Patients who have a surgery under general anesthesia
Anesthesia scheme for re-operation | up to 5 years
  Total intravenous anesthesia, inhalational anesthesia or combined anesthesia
Radiotherapy rate for any cancer | up to 5 years
  Patients have radiotherapy for any cancer
Chemotherapy rate for any cancer | up to 5 years
  Patients have chemotherapy for any cancer
Circulating tumor cells | up to 5 years
  Blood will be drawn preoperatively (at least 24 hours before surgery), prior to anesthesia induction, immediately postoperatively, 24 hours postoperatively, and at postoperative appointments for testing circulating tumor cells
Concentration of cytokines | up to 5 years
  Blood will be drawn preoperatively (at least 24 hours before surgery), prior to anesthesia induction, immediately postoperatively, 24 hours postoperatively, and at postoperative appointments for testing IL, TNF-α, IFN-γ and GCSF
Colorectal cancer antibodies | up to 5 years
  Blood will be drawn preoperatively (at least 24 hours before surgery), prior to anesthesia induction, immediately postoperatively, 24 hours postoperatively, and at postoperative appointments for testing CEA, CA199, GP87 and TPA.

OTHER OUTCOMES:
Re-operation during hospitalization | From end of colorectal cancer resection surgery to discharge, up to one month
  Patients receive a reoperation for any reason during hospitalization
Days of hospitalization | From end of colorectal cancer resection surgery to discharge, up to one month
  The duration of patients stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, MD, PhD, Study Chair — Department of Anesthesiology, West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Department of Anesthesiology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
All the study outcomes

REFERENCES:
- [Background] Sofra M, Fei PC, Fabrizi L, Marcelli ME, Claroni C, Gallucci M, Ensoli F, Forastiere E. Immunomodulatory effects of total intravenous and balanced inhalation anesthesia in patients with bladder cancer undergoing elective radical cystectomy: preliminary results. J Exp Clin Cancer Res. 2013 Feb 3;32(1):6. doi: 10.1186/1756-9966-32-6. PMID 23374147
- [Background] Qiao Y, Feng H, Zhao T, Yan H, Zhang H, Zhao X. Postoperative cognitive dysfunction after inhalational anesthesia in elderly patients undergoing major surgery: the influence of anesthetic technique, cerebral injury and systemic inflammation. BMC Anesthesiol. 2015 Oct 23;15:154. doi: 10.1186/s12871-015-0130-9. PMID 26497059
- [Background] Moller Petrun A, Kamenik M. Bispectral index-guided induction of general anaesthesia in patients undergoing major abdominal surgery using propofol or etomidate: a double-blind, randomized, clinical trial. Br J Anaesth. 2013 Mar;110(3):388-96. doi: 10.1093/bja/aes416. Epub 2012 Nov 19. PMID 23166149
- [Background] Jaura AI, Flood G, Gallagher HC, Buggy DJ. Differential effects of serum from patients administered distinct anaesthetic techniques on apoptosis in breast cancer cells in vitro: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i63-7. doi: 10.1093/bja/aet581. Epub 2014 Jul 9. PMID 25009197
- [Background] Buckley A, McQuaid S, Johnson P, Buggy DJ. Effect of anaesthetic technique on the natural killer cell anti-tumour activity of serum from women undergoing breast cancer surgery: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i56-62. doi: 10.1093/bja/aeu200. Epub 2014 Jul 9. PMID 25009196
- [Background] Wigmore TJ, Mohammed K, Jhanji S. Long-term Survival for Patients Undergoing Volatile versus IV Anesthesia for Cancer Surgery: A Retrospective Analysis. Anesthesiology. 2016 Jan;124(1):69-79. doi: 10.1097/ALN.0000000000000936. PMID 26556730
- [Background] Woo JH, Baik HJ, Kim CH, Chung RK, Kim DY, Lee GY, Chun EH. Effect of Propofol and Desflurane on Immune Cell Populations in Breast Cancer Patients: A Randomized Trial. J Korean Med Sci. 2015 Oct;30(10):1503-8. doi: 10.3346/jkms.2015.30.10.1503. Epub 2015 Sep 12. PMID 26425050
- [Background] Bayliss DA, Barrett PQ. Emerging roles for two-pore-domain potassium channels and their potential therapeutic impact. Trends Pharmacol Sci. 2008 Nov;29(11):566-75. doi: 10.1016/j.tips.2008.07.013. Epub 2008 Sep 25. PMID 18823665
- [Background] Pei L, Tan G, Wang L, Guo W, Xiao B, Gao X, Wang L, Li H, Xu Z, Zhang X, Zhao J, Yi J, Huang Y. Comparison of combined general-epidural anesthesia with general anesthesia effects on survival and cancer recurrence: a meta-analysis of retrospective and prospective studies. PLoS One. 2014 Dec 30;9(12):e114667. doi: 10.1371/journal.pone.0114667. eCollection 2014. PMID 25548913
- [Background] Shi C, Thum C, Zhang Q, Tu W, Pelaz B, Parak WJ, Zhang Y, Schneider M. Inhibition of the cancer-associated TASK 3 channels by magnetically induced thermal release of Tetrandrine from a polymeric drug carrier. J Control Release. 2016 Sep 10;237:50-60. doi: 10.1016/j.jconrel.2016.06.044. Epub 2016 Jul 1. PMID 27374629